CLINICAL TRIAL: NCT03423498
Title: The Possibility of the Activation of the Abductor Hallucis Muscle as a Result of the Toe-spread-out Exercise in Patients With Hallux Valgus and in People Without the Deformity: Clinical Trial.
Brief Title: The Toe-spread-out Exercise in Patients With Hallux Valgus and Without the Deformity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Małgorzata Eliks, Assistant, MSc, Poznan University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 886/15
Record Dates: First submitted 2018-01-21; First posted 2018-02-06 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Hallux Valgus
Keywords: hallux valgus,; toe-spread-out exercise; abductor hallucis muscle; surface electromyography
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- groups with toe-spread-out exercise (Experimental): This arm included individuals with hallux valgus (research group A) and without deformation (research group B), who were patients of Department of Rehabilitation, Poznan University of Medical Sciences. They performed the toe-spread-out exercises for 14 days and were examined twice: before and after exercises. The examination of participants included a surface electromyography, electroneurography and goniometer tests to measure the range of motion in the hallux joints.
  Interventions: Other: toe-spread-out exercise
- control group (No Intervention): This arm included individuals with hallux valgus deformity from the control group which did not undergo any therapy of hallux. They were patients of Department of Rehabilitation as well. These participants were examined twice at an interval of 14 days in the same way as the patients from experimental arm.

INTERVENTIONS:
Other: toe-spread-out exercise — The therapeutic intervention lasted 14 days and focused on doing the TSO exercise. This exercise was performed unilaterally under the supervision of a qualified physiotherapist. The starting position of the TSO exercise was the sitting position with the knee joint and hip bent at 90 degrees. The exercise consisted of 3 consecutive phases: dorsiflexion of the toes keeping the metatarsal heads and the heel on the ground, moving the fifth toe down and in a lateral direction, moving the big toe down and abduction. The final position needs to be maintained for 5 seconds. The whole sequence was repeated 200 times a day.
  Arms: groups with toe-spread-out exercise

SUMMARY:
The effectiveness of conservative treatment of hallux valgus deformity has not been sufficiently explored yet. The aim of this study was to assess the effect of the toe-spread-out exercise on the amplitude and frequency pattern in a surface electromyographic examination in patients with hallux valgus and in people without the deformity. An additional objective is the assessment of nerve conduction in an electroneurography and the assessment of range of motion in a clinical examination.

DETAILED DESCRIPTION:
The study design was based on an interventional model (clinical trial). The participants were assigned to two research groups (A - with diagnosis of hallux valgus and B- without the deformity) that received therapeutic intervention of the TSO exercise performed unilaterally. The unexercised feet could have caused a synergistic effect and falsified the results, thus the unexercised feet were excluded from the control group. Nevertheless, a small control group which did not undergo any hallux therapy was created to check if any changes in analysed parameters are actually related to the intervention. These control group patients were examined twice at an interval of 14 days.

The hallux deformities were assessed on the basis of X-ray images taken in weight-bearing conditions, in a standing position in the anterior-posterior projection. On all X-rays the hallux valgus angles (HVA) and the first intermetatarsal angles (FIA) were designated and measured by one radiologist.

Additionally, each patient with hallux valgus was assessed according to the Hallux Metatarsophalangeal-Interphalangeal scale (HMP-IP scale) developed by the AOFAS (American Orthopaedic Foot and Ankle Society).

The effects of the exercises were assessed using a comparison of the outcomes of two examinations: before and after therapy (research group A and B). For this purpose, a surface electromyographic examination (sEMG) recorded from the abductor hallucis (AbdH) muscle was performed. The following parameters of electromyography were analysed in three phases of TSO exercise: amplitude and frequency pattern. Additionally, the motor fibres of the tibial nerve and the sensory fibres of the sural nerve function in electroneurographic examination (ENG) and range of motion of hallux using goniometer were assessed.

The sEMG recorded from the AbdH muscle and the ENG were performed with the use of the KeyPoint System (Medtronic A/S, Skovlunde, Denmark) and appropriate to the type of neurophysiological studies and set of electrodes (surface electrodes, bipolar stimulating electrode, and grounding electrode).

For the analysis of the bioelectrical activity of the AbdH the standard disposable Ag/AgCl surface electrodes with an active surface of 5mm2 were applied. The active electrode (cathode) was located on the belly muscle and the reference electrode (anode) was attached 3 cm distally from the active electrode. For the purpose of the sEMG examinations, the time base on 80ms/D and sensitivity of the recording of 0.5mV/D were set. 10kHz upper and 20Hz lower filters of the recorder amplifier were used.

The sEMG recordings were performed during three phases of the TSO exercise. The following parameters were analysed: amplitude of motor unit action potential (MUAP) measured in mV, and the frequency pattern of the MUAP recruitment of AbdH muscle activity. The sEMG tests with maintaining each phase of the TSO exercise were performed three times in order to obtain more objective results. The first test was treated as a training trial. The other two were taken into account to assess the amplitude and the frequency pattern. Only the trial with the highest amplitude and the most interference pattern was analysed as the result of the most effective recruitment of the MUAPs. The minimal and maximal amplitude values were automatically measured by the KeyPoint System after the marking of the MUAP amplitude peaks. An 'on-line' evaluation of the frequency of the MUAP recruitment during a maximal muscle contraction was a subjective visual assessment made by one experienced neurophysiologist. It was based on the following classification patterns presented by Buchthal et al. and by Stalberg and Falck: interference, intermediate, poor, and straight.

In the ENG the following parameters of the CMAP (compound muscle action potential) from the tibial nerve and of the SNAP (sensory nerve action potential) from the sural nerve were analysed: amplitude (measured from a negative inflection to the baseline in mV or in µV), latency (measured in ms) and conduction velocity (measured in m/s). During the ENG the time base on 5ms/D and sensitivity of the recordings on 2mV/D were set. 10Hz upper and 10kHz lower filters of the recorder amplifier were used. In order to record the compound muscle action potentials (CMAP) evoked from the AbdH muscle, the same location of surface electrodes as in the EMG was used. The electrical stimulation of the tibial nerve was applied in two points: below the medial malleolus and in the popliteal fossa. The ground electrode was located in the plantar part of the foot. Single rectangular stimuli with duration of 0.2ms were delivered via bipolar electrode at 1Hz frequency while their intensity ranged from 30mA to the value evoking the supramaximal CMAP. For recordings of SNAP from the sural nerve antidromic and repetitive electrical stimulation with an intensity of 20 mA was required. Recording electrodes were placed near the lateral malleolus while the stimulation point was 15 cm proximally at the external border of the Achilles tendon.

A clinical examination with the use of a goniometer was performed in the supine position of the patient. The investigator measured the range of the motion of the plantar and dorsal flexion in the first metatarsophalangeal joint and plantar flexion in the hallux interphalangeal joint.

ELIGIBILITY:
Inclusion Criteria:

* for patients with hallux valgus (research group A and control group): "B", "C" or "D" score in the Manchester scale, hallux valgus angle above 15° • for healthy volunteers (research group B) "A" score in the Manchester scale, hallux valgus angle equal or lower than 15°

Exclusion Criteria:

* for all groups: a serious injury or a history of lower limb surgery, presence of pain from a disc disease on the background of the disco-radicular conflict (based on the ENG study), neuropathy, myopathy, rheumatoid arthritis, psoriatic arthritis, connective tissue diseases, a history of strokes or other neurological diseases.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-10-20 (Actual); Primary Completion 2017-09-10 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Evaluation of changes in amplitude of motor unit action potential (MUAP) | 2 weeks (14 days)
  The amplitude of motor unit action potential (MUAP) recorded from the abductor hallucis muscle in three phases of exercise and measured in mV

SECONDARY OUTCOMES:
Evaluation of changes in frequency pattern of abductor hallucis muscle activity | 2 weeks (14 days)
  The frequency pattern of the MUAP recruitment of abductor hallucis muscle activity based on the following classification patterns presented by Buchthal et al. and by Stalberg and Falck: interference (IF), intermediate (IM), poor (P) and straight (S).

OTHER OUTCOMES:
Evaluation of changes in amplitude of the CMAP (compound muscle action potential) from the tibial nerve and of the SNAP (sensory nerve action potential) from the sural nerve | 2 weeks (14 days)
  The amplitude measured from a negative inflection to the baseline in mV.
Evaluation of changes in latency of the CMAP (compound muscle action potential) from the tibial nerve and of the SNAP (sensory nerve action potential) from the sural nerve | 2 weeks (14 days)
  The latency measured in ms.
Evaluation of changes in conduction velocity of the CMAP (compound muscle action potential) from the tibial nerve and of the SNAP (sensory nerve action potential) from the sural nerve | Time frame: 2 weeks (14 days)
  The conduction velocity measured in m/s.

CONTACTS AND LOCATIONS:
Overall Officials: Przemysław Lisiński, MD, PhD, Study Director — Poznan University of Medical Sciences; Kamila Mortka, Msc, Principal Investigator — Poznan University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arinci Incel N, Genc H, Erdem HR, Yorgancioglu ZR. Muscle imbalance in hallux valgus: an electromyographic study. Am J Phys Med Rehabil. 2003 May;82(5):345-9. doi: 10.1097/01.PHM.0000064718.24109.26. PMID 12704272
- [Background] Hoffmeyer P, Cox JN, Blanc Y, Meyer JM, Taillard W. Muscle in hallux valgus. Clin Orthop Relat Res. 1988 Jul;(232):112-8. PMID 3383479
- [Background] Kim MH, Kwon OY, Kim SH, Jung DY. Comparison of muscle activities of abductor hallucis and adductor hallucis between the short foot and toe-spread-out exercises in subjects with mild hallux valgus. J Back Musculoskelet Rehabil. 2013;26(2):163-8. doi: 10.3233/BMR-2012-00363. PMID 23640317
- [Background] Kim MH, Yi CH, Weon JH, Cynn HS, Jung DY, Kwon OY. Effect of toe-spread-out exercise on hallux valgus angle and cross-sectional area of abductor hallucis muscle in subjects with hallux valgus. J Phys Ther Sci. 2015 Apr;27(4):1019-22. doi: 10.1589/jpts.27.1019. Epub 2015 Apr 30. PMID 25995546
- [Background] BUCHTHAL F, PINELL P, ROSENFALCK P. Action potential parameters in normal human muscle and their physiological determinants. Acta Physiol Scand. 1954 Nov;32(2-3):219-29. doi: 10.1111/j.1748-1716.1954.tb01168.x. No abstract available. PMID 13228110
- [Background] Stalberg E, Falck B. The role of electromyography in neurology. Electroencephalogr Clin Neurophysiol. 1997 Dec;103(6):579-98. doi: 10.1016/s0013-4694(97)00138-7. PMID 9546485